CLINICAL TRIAL: NCT00399399
Title: CHUSPAN SCS BP Treatment of Churg-Strauss Syndrome Without Poor-Prognosis Factors: a Prospective Randomized Study in 72 Patients.
Brief Title: CHUSPAN SCS BP Treatment of Churg-Strauss Syndrome Without Poor-Prognosis Factors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 95.067
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2006-11

CONDITIONS: Churg-Strauss Syndrome
Keywords: Churg-Strauss; Vasculitis; Therapy; Cyclophosphamide; Azathioprine
MeSH Terms: conditions — Churg-Strauss Syndrome; Vasculitis | interventions — Azathioprine; Cyclophosphamide

INTERVENTIONS:
Drug: azathioprine
Drug: cyclophosphamide

SUMMARY:
To assess the efficacy of systemic corticosteroids alone as first-line treatment of Churg-Strauss syndrome without poor-prognosis factors as defined by the five-factor score (FFS=0), and to compare the efficacy and safety of azathioprine vs pulse cyclophosphamide as adjunctive immunosuppressive therapy to treat failure or relapse

DETAILED DESCRIPTION:
All patients initially treated with systemic corticosteroids alone: optional IV methylprednisolone pulse (15 mg/kg) at treatment start followed by oral prednisone (1 mg/kg/day) according to a tapering schedule. Treating physicians allowed to treat minor relapses with corticosteroids without referring the patient for randomization, as long as the prednisone dose did not exceed 0.5 mg/kg for 1 month.

Patients in whom prednisone doses could not be tapered below 20 mg, those who failed to enter remission and those who relapsed were randomized to receive either 6 months of oral azathioprine (2mg/kg/day) or 6 cyclophosphamide pulses (0.6g/m2 D1, D15, D30 then every month)

ELIGIBILITY:
Inclusion Criteria:

* Men and women with newly diagnosed Churg-Strauss syndrome;
* absence of poor prognostic factors as defined by the five-factor score (serum creatinine > 140 μmol/l or 1.58 mg/dl, proteinuria > 1 g/day, severe gastrointestinal tract involvement, specific cardiomyopathy and/or central nervous system involvement;
* written informed consent.

Exclusion Criteria:

* age < 15 years, previously treated Churg-Strauss syndrome;
* history of cancer;
* pregnant or breast-feeding women;
* psychiatric disorders that might compromise compliance with therapy;
* contraindication to study drug;
* other ongoing therapeutic trial;
* concomitant viral hepatitis B or C or human immunodeficiency virus (HIV) infection

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72
Dates: Start 1996-07

PRIMARY OUTCOMES:
Number of events (failures, relapses and/or deaths) occurring in each group, defining the disease-free survival rate, measured at study end (mean follow-up of 5 years)

SECONDARY OUTCOMES:
Overall survival, relapse rate and adverse events, measured at study end (mean follow-up of 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Cordier, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Camillo Ribi, Geneva, Switzerland

REFERENCES:
- [Derived] Samson M, Puechal X, Devilliers H, Ribi C, Cohen P, Bienvenu B, Terrier B, Pagnoux C, Mouthon L, Guillevin L; French Vasculitis Study Group (FVSG). Mononeuritis multiplex predicts the need for immunosuppressive or immunomodulatory drugs for EGPA, PAN and MPA patients without poor-prognosis factors. Autoimmun Rev. 2014 Sep;13(9):945-53. doi: 10.1016/j.autrev.2014.08.002. Epub 2014 Aug 19. PMID 25153486
- [Derived] Samson M, Puechal X, Devilliers H, Ribi C, Cohen P, Stern M, Pagnoux C, Mouthon L, Guillevin L; French Vasculitis Study Group. Long-term outcomes of 118 patients with eosinophilic granulomatosis with polyangiitis (Churg-Strauss syndrome) enrolled in two prospective trials. J Autoimmun. 2013 Jun;43:60-9. doi: 10.1016/j.jaut.2013.03.003. Epub 2013 Apr 13. PMID 23590801
- [Derived] Ribi C, Cohen P, Pagnoux C, Mahr A, Arene JP, Lauque D, Puechal X, Letellier P, Delaval P, Cordier JF, Guillevin L; French Vasculitis Study Group. Treatment of Churg-Strauss syndrome without poor-prognosis factors: a multicenter, prospective, randomized, open-label study of seventy-two patients. Arthritis Rheum. 2008 Feb;58(2):586-94. doi: 10.1002/art.23198. PMID 18240234